CLINICAL TRIAL: NCT00563823
Title: A Phase II Study to Evaluate the Efficacy and Safety of PTK787 in Patients With Metastatic Cutaneous Melanoma
Brief Title: Vatalanib in Treating Patients With Metastatic Cutaneous Melanoma That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CRCA-CCTC-CAMEL02; CDR0000576458 (Registry Identifier: PDQ (Physician Data Query)); EU-20787; EUDRACT-2005-004710-33; CCLG-Camel-02; ISRCTN00191981 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register))
Record Dates: First submitted 2007-11-22; First posted 2007-11-26 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-04

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — vatalanib

INTERVENTIONS:
Drug: vatalanib

SUMMARY:
RATIONALE: Vatalanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well vatalanib works in treating patients with metastatic cutaneous melanoma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate in patients with unresectable metastatic cutaneous melanoma treated with vatalanib.

Secondary

* To determine the time to progression in these patients.
* To determine the 6-month and 1-year survival of these patients.
* To determine the overall survival of these patients.
* To determine the safety and toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral vatalanib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed at 8 weeks and then periodically thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic cutaneous melanoma

  * Unresectable disease
* Measurable disease, defined as ≥ 1 bidimensionally measurable lesion by clinical or radiological techniques (i.e., chest x-ray, CT scan, or conventional MRI scan) using RECIST criteria
* No history or presence of CNS disease (i.e., primary brain tumor, malignant seizures, clinically symptomatic CNS metastases, or carcinomatous meningitis)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Bilirubin ≤ 1.5 x upper limit of normal (ULN)
* Alkaline phosphatase ≤ 3 x ULN (≤ 5 if liver metastases are present)
* Transaminases ≤ 3 x ULN (≤ 5 if liver metastases are present)
* Creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min
* Total urinary protein ≤ 500 mg by 24-hour urine collection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No history of other malignant disease except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No other serious or uncontrolled illness which, in the opinion of the investigator, precludes study entry
* No medical or psychiatric condition that precludes giving informed consent
* No history of renal disease (e.g., glomerulonephritis) or renal vascular disease
* No acute or chronic active liver disease (e.g., hepatitis or cirrhosis)
* No concurrent severe and/or uncontrolled medical conditions that would compromise participation in the study, including any of the following:

  * Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
  * Unstable angina pectoris
  * Symptomatic congestive heart failure
  * Myocardial infarction within the past 6 months
  * Serious uncontrolled cardiac arrhythmia
  * Uncontrolled diabetes
  * Active or uncontrolled infection
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of vatalanib including, but not limited to, any of the following conditions:

  * Ulcerative disease
  * Uncontrolled nausea
  * Vomiting
  * Diarrhea which might result in malabsorption
  * Any known malabsorption syndrome
  * Bowel obstruction
  * Inability to swallow the capsules/tablets

PRIOR CONCURRENT THERAPY:

* Recovered from all prior therapy
* Prior adjuvant therapy allowed
* Prior radiotherapy allowed

  * Measurable target lesions must not have been irradiated
* No more than one line of prior systemic therapy for advanced melanoma
* More than 4 weeks since prior chemotherapy, immunotherapy, or investigational agent
* More than 2 weeks since prior surgery
* No concurrent warfarin or other similar oral anticoagulants that are metabolized by the cytochrome p450 system

  * Concurrent heparin allowed
* Concurrent radiotherapy for symptomatic disease is allowed, provided the lesions being irradiated contribute ≤ 20% of the sum of the longest diameter for all target lesions being used to determine response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Response rate as assessed by RECIST every 8 weeks

SECONDARY OUTCOMES:
Time to progression
Survival at 6 months and 1 year
Overall survival
Toxicity as assessed by NCI CTCAE v3.0 at 2 weeks and then every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, PhD, FRCP, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge, England
  - Leicester Royal Infirmary, Leicester, England

REFERENCES:
- [Result] Cook N, Basu B, Biswas S, Kareclas P, Mann C, Palmer C, Thomas A, Nicholson S, Morgan B, Lomas D, Sirohi B, Mander AP, Middleton M, Corrie PG. A phase 2 study of vatalanib in metastatic melanoma patients. Eur J Cancer. 2010 Oct;46(15):2671-3. doi: 10.1016/j.ejca.2010.07.014. Epub 2010 Aug 25. PMID 20800475